CLINICAL TRIAL: NCT00163033
Title: Phase I Study to Evaluate the Safety, Tolerability, PK and Pharmacodynamics of 3 Dosages of Estetrol, the Lowest Dose of 2 mg Estetrol Compared With 2 mg of E2, After Daily Oral Administration for 28 Days in Healthy Postmenopausal Women
Brief Title: Study to Evaluate 3 Dosages of Estetrol After 28 Days Administration in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pantarhei Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR3054
Record Dates: First submitted 2005-09-12; First posted 2005-09-13 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: phase I study
MeSH Terms: interventions — Estetrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: estetrol

SUMMARY:
Estetrol is a natural compound that is produced by the fetus during fetal life and circulates in the unborn child and the mother. It is an estrogenic compound. In this study the safety and tolerability of 28 days of the oral administration of estetrol in healthy postmenopausal women are investigated. In addition, the pharmacokinetics and some pharmacodynamic parameters are studied. The lowest dose of 2 mg estetrol is directly compared with 2 mg estradiol.

DETAILED DESCRIPTION:
This is a partly randomized open-label study in healthy postmenopausal women. Groups are treated in the following sequence: first a 2 mg estetrol group together with a 2 mg estradiol group. When the dose of 2 mg estetrol is safe and the tolerability is good, a next higher dose group of estetrol will start, possibly followed by two next higher dose groups if the previous dose group is safe and the tolerability is good.

The primary objective of this study is to investigate the safety and tolerability of estetrol during multiple dosing for 28 days. Furthermore steady state pharmacokinetics and some pharmacodynamic parameters of estetrol will be investigated. In addition, the pharmacokinetics and pharmacodynamic effects of the 2 mg estetrol group will be compared with those of the 2 mg estradiol group.

In each group 5 postmenopausal women will be included with > 50 hot flushes per week and 5 postmenopausal women with < 10 hot flushes per week. These criteria are set to get a more homologous composition in each group.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women not older than 70 years of age at the time of screening (menopause defined as ≥ 6 months amenorrhea with serum follicle-stimulating hormone [FSH] levels ≥ 40 IU/L and serum E2 < 73 pmol/L).
* Body mass index 18-30 kg/m2 inclusive.
* Good physical and mental health, as judged by the Investigator, determined by medical history, physical examination, clinical laboratory values, vital signs, and electrocardiogram (ECG) recording.
* Willing to give written informed consent.
* Either > 50 hot flushes per week or < 10 hot flushes per week

Exclusion Criteria:

* Clinically significant abnormal results of routine hematology, serum biochemistry, urinalysis, and/or ECG in the opinion of the Investigator at screening.
* Clinically significant abnormal mammogram (presence of any non-cystic mass) within one year before study start.
* Clinically significant abnormalities of the uterus and/or ovaries detected by examination and/or ultrasound (non-physiological ovarian mass or significant uterine pathology or an endometrium greater than 6 mm).
* A cervical smear with clinically relevant abnormal cytology within one year before study start.
* Previous use of estrogen/progestogen within:

  * 6 months for depot preparations.
  * 8 weeks for oral preparations or progestogen containing intrauterine device (IUD).
  * 4 weeks for transdermal preparations.
* Use of hormone containing implant at any time.
* Contraindications for using steroids:

  * A history of, or existing thromboembolic, cardiovascular, or cerebrovascular disorder.
  * A history of, or existing conditions predisposing to, or being prodrome of, a thrombosis.
  * A known defect in the blood coagulation system (e.g. deficiencies in antithrombin-III [AT-III], protein C, S, and activated protein C [APC] resistance).
  * A medical history positive for the presence of more than one risk factor for vascular disease (e.g. dyslipoproteinemia; diabetes mellitus; hyperhomocysteinemia; systemic lupus erythematosus; chronic inflammatory bowel disease; smoking; venous thromboembolism in sibling or parent below the age of 50, or arterial disease in sibling or parent below the age of 30-35).
  * Hypertension, i.e. systolic blood pressure >160 mm Hg and/or diastolic blood pressure >100 mm Hg.
  * Disturbance of liver function: cholestatic jaundice, a history of jaundice in pregnancy or jaundice due to previous estrogen use, Rotor syndrome and Dubin-Johnson syndrome.
  * Known or suspected estrogen-dependent tumors or endometrial hyperplasia
  * Undiagnosed vaginal bleeding.
  * Porphyria.
  * A history during pregnancy or previous estrogen use of severe pruritus, herpes gestationis, or deterioration of otosclerosis.
* Any medication (including over-the-counter [OTC] products) from 14 days prior to the day of dosing except for occasional non-steroidal anti-inflammatory drugs (NSAID; e.g. ibuprofen); paracetamol is not permitted.
* Any enzyme affecting drugs from 30 days prior to Day 1 and the use of griseofulvin, primidone, oxcarbazepine, topiramate, felbamate, or herbal remedies containing hypericum perforatum (St. John's wort).
* Presence of significant allergies or other serious diseases.
* Smoking more than 10 cigarettes or equivalent per day.
* Administration of investigational drugs within 3 months before start of study medication.
* A history of (within 12 months) alcohol or drug abuse.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-06; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
safety of estetrol
tolerability of estetrol

SECONDARY OUTCOMES:
steady state pharmacokinetics of estetrol
pharmacodynamic effects of estetrol
to compare the pharmacokinetics and pharmacodynamic effects of 2 mg estetrol with 2 mg estradiol
to investigate the effect on the number of hot flushes and sweating of 2 mg estetrol compared with 2 mg estradiol

CONTACTS AND LOCATIONS:
Overall Officials: Herjan Coelingh Bennink, MD, PhD, Study Director — Pantarhei Bioscience
Locations (1):
- Kendle Clinical Pharmacology Unit, Utrecht, Utrecht, Netherlands